CLINICAL TRIAL: NCT06769100
Title: The Effects of Ketone Monoester Intake on Postprandial Myofibrillar Protein Synthesis Rates in Young Adults During Recovery Following an Acute Bout of Resistance Exercise
Brief Title: Exogenous Ketosis and Muscle Protein Synthesis During Exercise Recovery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University (Other)
Responsible Party: Principal Investigator, Tyler Churchward-Venne, Associate Professor, McGill University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: A00-M15-24A
Record Dates: First submitted 2025-01-06; First posted 2025-01-10 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Ketosis; Muscle Protein Synthesis; Dietary Proteins; Resistance Exercise
Keywords: Ketosis; Regulation of Muscle Protein Synthesis; Resistance Exercise; Post-Exercise Recovery; Whey Protein
MeSH Terms: conditions — Ketosis | interventions — Whey Proteins; Resistance Training

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants, Investigators and Outcome Accessors will be blinded to the intervention and control drinks. The drinks will be flavor matched and provided in an opaque bottle. An individual not involved with the study data collection, analysis and interpretation will be designated as a study blinder and randomizer.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Ketone Monoester (KET) (Experimental): Ketone monoester supplement (R)-3-hydroxybutyl (R)-3-hydroxybutyrate based on participants' body weight (0.36g/kg body weight).
  Interventions: Dietary Supplement: Ketone Monoester (KET); Other: Resistance exercise
- Ketone Monoester + Whey Protein (KET+PRO) (Experimental): Ketone monoester supplement (R)-3-hydroxybutyl (R)-3-hydroxybutyrate based on participants' body weight (0.36g/kg body weight) and 25g of whey protein.
  Interventions: Dietary Supplement: Ketone Monoester + Whey Protein (KET+PRO); Other: Resistance exercise
- Whey Protein (PRO) (Experimental): 25g of whey protein.
  Interventions: Dietary Supplement: Whey Protein (PRO); Other: Resistance exercise
- Placebo drink (CON) (Placebo Comparator): Flavoured water.
  Interventions: Dietary Supplement: Flavour matched placebo (CON); Other: Resistance exercise

INTERVENTIONS:
Dietary Supplement: Ketone Monoester (KET) — - Ketone monoester supplement (R)-3-hydroxybutyl (R)-3-hydroxybutyrate based on participants' body weight (0.36g/kg body weight). The ketone brand name: delta G Oxford Ketone Ester
  Arms: Ketone Monoester (KET)
Dietary Supplement: Ketone Monoester + Whey Protein (KET+PRO) — * Ketone monoester supplement (R)-3-hydroxybutyl (R)-3-hydroxybutyrate based on participants' body weight (0.36g/kg body weight)
  * 25g Whey Protein
  * L-[ring-2H5]-phenylalanine tracer (enriched to 4%)
  Arms: Ketone Monoester + Whey Protein (KET+PRO)
Dietary Supplement: Whey Protein (PRO) — * 25g Whey Protein
  * L-[ring-2H5]-phenylalanine tracer (enriched to 4%)
  Arms: Whey Protein (PRO)
Dietary Supplement: Flavour matched placebo (CON) — - Flavoured water (non-caloric bitter + citrus flavours)
  Arms: Placebo drink (CON)
Other: Resistance exercise — - 8 sets of 10 reps at 90% of 10- repetition maximum (10-RM) of unilateral leg extension with 90 seconds rest in between sets.

SUMMARY:
An acute bout of resistance exercise stimulates muscle protein synthesis (MPS) rates for up to 24-48 hours, supporting muscle growth and repair. To optimize the anabolic effects of resistance exercise, the provision of dietary amino acids (i.e., proteins) is essential. Dietary protein intake provides the body with necessary amounts of essential and non-essential amino acids, which represent the building blocks for muscle proteins, enhancing anabolic muscle growth. The ingestion of dietary protein, such as whey protein, is well established to stimulate an increase in the rate of protein synthesis in skeletal muscle following resistance exercise. Research has demonstrated a dose-dependent relationship between protein intake and MPS rate, with 25 grams being the optimal dose to maximally stimulate MPS rates in younger adults with excess protein oxidized as a fuel source.

Determining whether this maximally stimulated MPS response can be further heightened during post-exercise recovery using non-protein dietary factors is yet to be explored. Recently, it has been shown that novel orally ingested ketone body supplements can stimulate MPS rates in younger adults at rest.

Ketone bodies (β-OHB) are lipid- derived molecules normally produced under conditions of glucose deprivation (i.e., fasting/starvation, or a low carbohydrate 'ketogenic' diet). However, these orally ingested ketone supplements rapidly increase blood ketone levels without the need for dietary restriction6. In vitro research showed that the combination of leucine and ketone bodies stimulated a 2-fold increase in MPS, compared to the leucine group alone, indicating synergistic effects of protein and ketone bodies on MPS. However, the effect of ketone supplementation, with and without dietary protein co-ingestion, on MPS rate during post-exercise recovery is yet to be investigated. If ketone bodies can amplify the anabolic response to dietary protein, they may provide a novel approach to maximizing muscle adaptation during post-exercise recovery.

Therefore, the purpose of this study is to evaluate the effects of ketone monoester intake on postprandial muscle protein synthesis rates when consumed alone and when co-ingested with an optimal dose (25 g) of whey protein during recovery after resistance exercise compared to 1) an optimal dose of whey protein (25 g), and 2) a control flavored water. It is hypothesized that muscle protein synthesis rates will be stimulated following the ingestion of the ketone body beverage. Further, muscle protein synthesis rates will be further enhanced when the ketone-containing beverage and an optimal dose are taken together.

DETAILED DESCRIPTION:
A parallel group design will be used for this randomized double-blind, placebo-controlled study in healthy adults to investigate the effects of ketone monoester on myofibrillar protein synthesis rates during post-exercise recovery. There are 4 groups in this trial, including one ketone group (0.36g/kg body weight) (KET), one protein group (25 g whey protein) (PRO), a combination of ketone and protein (KET+PRO), and a placebo group (flavoured water) (CON). A total of 48 participants will be enrolled in this trial (n=12 per group).

The study will include a screening visit (visit 1), 10-repetition maximum (10-RM) testing (visit 2), where participants' 10-RM will be determined for the exercise protocol, and the experimental trial (visit 3).

During the experimental trials, participants will arrive to the laboratory in a fasted state, and a prime dose of the L-[ring-2H5]-phenylalanine will be administered followed by a continuous infusion at a rate 0.05 μmol/kg of body weight/min. Then, participants will perform a unilateral lower-body resistance exercise, consisting of 8 sets of 10 reps of unilateral leg extension at 90% of their 10-RM with 90 seconds rest in between sets. Following exercise, the nutritional treatment will be administered.

Arterialized blood will be collected at baseline and 13 postprandial timepoints across 9 hours for plasma amino acid, glucose, and insulin quantitation.

Additionally, changes in capillary blood β-HB concentration will be assessed throughout the trial by collecting capillary blood samples at baseline and 10 postprandial timepoints. Finally, muscle biopsy samples from both the exercised leg and the rested leg will be collected prior to beverage intake and at the 5-hour mark of the postprandial post-recovery period to assess myofibrillar protein synthesis rates.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult female or male participants who are 18-40 years of age (inclusive) BMI >18.5 and <30.0 kg/m2
* Moderately active (i.e., ≥ 1 session of lower-body weightlifting /week for the previous 2 months).
* Has maintained stable use of medication and supplements (which are not limited by the exclusion criteria), stable dietary and lifestyle habits, and stable body weight, for the last 3 months prior to screening and agree to maintain them throughout the study.
* Be willing to entirely avoid alcohol consumption 48hr prior to the experimental test day.
* Willing and able to agree to the requirements and restrictions of this study, be willing to give voluntary consent, be able to understand and read the questionnaires, and carry out all study-related procedures.

Exclusion Criteria:

* Females who are lactating or pregnant
* Females using third-generation oral contraceptives (including: Desogen®, Ortho-Cept, Ortho-Cyclen, Ortho Tri-Cyclen) as these are known to affect protein metabolism in females.
* Individuals with metabolic disorders including: Type I or Type II diabetes
* Individuals with a history of thrombosis / cardiovascular disease
* Individuals who use of anticoagulants
* Individuals with musculoskeletal / orthopedic disorders
* Individuals with knee injuries (i.e., ACL injuries).
* Individuals who have used tobacco products within the last 6 months
* Individuals with a history of neuromuscular problems
* Chronic usage of medications known to modulate skeletal muscle metabolism (i.e. corticosteroids, hormone replacement therapy (HRT), and over-the-counter supplements including creatine monohydrate) in the last 6 months.
* Individuals with allergies to milk proteins (whey or casein).
* Individuals with lactose intolerance
* Individuals with Phenylketonuria (PKU)
* Previous participation in amino acid tracer studies.
* Adherence to a vegetarian or vegan diet
* Current use of ketone supplements or adherence to a ketogenic diet
* Individuals who train more than ≥ 5 sessions of lower-body weightlifting /week for the previous 4 months

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Cis males and Cis females
Enrollment: 48 (Estimated)
Dates: Start 2025-01-10 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Myofibrillar fractional synthesis rate | 0 - 5 hours in the postprandial period.
  Quantification of changes in basal myofibrillar fractional synthetic rate (%/hour) in the rested and exercised limbs.

SECONDARY OUTCOMES:
Time-course data for plasma enrichments (in moles percent excess) of L-[ring-2H5]-phenylalanine | Baseline, 3 hours pre-prandial, and 5 hours into the postprandial period.
  Changes in plasma-free L-[ring-2H5]-phenylalanine enrichment measured at 14 time points (t = -180, -120, -60, 0, 15, 30, 45, 60, 90, 120, 150, 180, 240, 300 minute).
Incremental area under the curve for total amino acid concentration | 3 hours pre-prandial to 5 hours postprandial
  Incremental area under the curve (iAUC) for plasma concentration of total amino acids (μmol/L) including: free leucine, isoleucine, valine, histidine, lysine, methionine, phenylalanine, threonine, tryptophan, arginine, glutamine, glycine, alanine, serine, glutamic acid, aspartic acid, asparagine, tyrosine, cysteine, proline (combined), measured at baseline and across the 3-hour pre-prandial period and 5-hour postprandial period.
Time-course data for total amino acid concentration | Baseline, 3 hours pre-prandial, and 5 hours into the postprandial period.
  Changes in plasma concentration of total amino acid concentration (μmol/L) including: free leucine, isoleucine, valine, histidine, lysine, methionine, phenylalanine, threonine, tryptophan, arginine, glutamine, glycine, alanine, serine, glutamic acid, aspartic acid, asparagine, tyrosine, cysteine, proline (combined), measured at 14 time points (t = -180, -120, -60, 0, 15, 30, 45, 60, 90, 120, 150, 180, 240, 300 minute).
Incremental area under the curve for essential amino acid concentration | 3 hours pre-prandial to 5 hours postprandial
  Incremental area under the curve (iAUC) for plasma essential amino acid concentration (μmol/L) including free leucine, isoleucine, valine, histidine, lysine, methionine, phenylalanine, threonine, tryptophan (combined), measured at baseline and across the 3-hour pre-prandial period and 5-hour postprandial period.
Time-course data for essential amino acid concentration | Baseline, 3 hours pre-prandial, and 5 hours into the postprandial period.
  Changes in plasma concentration of essential amino acid (μmol/L) including: free leucine, isoleucine, valine, histidine, lysine, methionine, phenylalanine, threonine, tryptophan (combined), measured at 14 time points (t = -180, -120, -60, 0, 15, 30, 45, 60, 90, 120, 150, 180, 240, 300 minute).
Incremental area under the curve for leucine concentration | 3 hours pre-prandial to 5 hours postprandial
  Incremental area under the curve (iAUC) for plasma leucine concentration (μmol/L) measured at baseline and across the 3-hour pre-prandial period and 5-hour postprandial period.
Time-course data for leucine concentration | Baseline, 3 hours pre-prandial, and 5 hours into the postprandial period.
  Changes in plasma concentration of leucine (μmol/L) measured at 14 time points (t = -180, -120, -60, 0, 15, 30, 45, 60, 90, 120, 150, 180, 240, 300 minute).
Incremental area under the curve for glucose concentration | 3 hours pre-prandial to 5 hours post-prandial
  Plasma glucose concentration (mmol/L) and its corresponding incremental area under the curve (iAUC), measured at baseline and across the 3-hour pre-prandial period and 5-hour postprandial period.
Time-course data for glucose concentration | Baseline, 3 hours pre-prandial, and 5 hours into the postprandial period.
  Changes in plasma concentration of glucose (mmol/L) measured at 14 time points (t = -180, -120, -60, 0, 15, 30, 45, 60, 90, 120, 150, 180, 240, 300 minute).
Incremental area under the curve for insulin concentration | 3 hours pre-prandial to 5 hours post-prandial
  Incremental area under the curve (iAUC) for plasma concentration of insulin (pmol/L), measured at baseline and across the 3-hour pre-prandial period and 5-hour postprandial period.
Time-course data for insulin concentration | Baseline, 3 hours pre-prandial, and 5 hours into the postprandial period.
  Changes in plasma concentration of insulin (pmol/L) measured at 14 time points (t = -180, -120, -60, 0, 15, 30, 45, 60, 90, 120, 150, 180, 240, 300 minute).
Incremental area under the curve for β-HB concentrations | 1 hour pre-prandial to 5 hours postprandial
  Capillary blood β-OHB concentration (mmol/L) and its corresponding incremental area under the curve (iAUC) measured during the pre-prandial period and postprandial period.
Time-course data for β-HB concentrations | 1 hour pre-prandial to 5 hours in the post-prandial period
  Changes in capillary blood β-OHB concentration (mmol/L) measured at 10 time points (t = -60, 0, 30, 60, 90, 120, 150, 180, 240, 300 minute).
Changes in the phosphorylation status of anabolic signaling molecules | 0 and 5 hours of the postprandial period.
  Western blot analysis will be used to measure the changes in the basal phosphorylation status of anabolic signaling molecules, including p-mTORC1 (Ser2448), p-p70S6K (Thr389), p-Akt (Ser473), p-4E-BP1 (Thr37/46), and p-rpS6 (Ser240/244), p-ERK1(Thr202/Tyr204), and p-ERK2 (Thr185/Tyr187), in the exercised and the rested limbs.

CONTACTS AND LOCATIONS:
Overall Officials: Tyler Churchward-Venne, PhD, Principal Investigator — Department of Kinesiology and Physical Education, McGill University
Locations (1):
- McGill University, Montreal, Quebec, Canada